CLINICAL TRIAL: NCT06284395
Title: Bortezomib, Thalidomide, and Dexamethasone Versus Thalidomide and Dexamethasone for Response Rates in Multiple Myeloma Patients: a Retrospective Study
Brief Title: Two Schemes Response in Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal investigator, Hospital General de Mexico
Other Study IDs: HGM1471-002/24
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Response, Acute Phase; Survivorship
Keywords: Multiple Myeloma; Bortezomib; Thalidomide; Acute Phase Response; Survival
MeSH Terms: conditions — Acute-Phase Reaction; Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Thalidomide 100mg-200mg PO daily alone or in combination with dexamethasone 40mg PO every 24 hours on days 1-4, 8-11 of each cycle.
  Interventions: Drug: Bortezomib
- Bortezomib Group: Bortezomib 1.3mg/m2 SC on days 1,4, 8,11 to the TD scheme for a total of 6 treatment cycles (VTD).
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3mg/m2 SC on days 1,4, 8,11 to the TD scheme for a total of 6 treatment cycles (14,15) (VTD)
  Other Names: Intervention Group

SUMMARY:
Retrospective study based on medical records of patients with multiple myeloma, eligible for stem cell transplantation, who received, first-line, the VTD or TD combination.

DETAILED DESCRIPTION:
The most current treatment of multiple myeloma is based on a combination of drugs, including immunomodulators, proteasome inhibitors, etc. The VTD (bortezomib, thalidomide, and dexamethasone) and TD (thalidomide and dexamethasone) regimens are commonly used as a first-line treatment due to limited resources. The study aimed to compare the proportion of favorable responses, survival, and time to the next treatment between two different treatment approaches. The investigators designed a retrospective study based on medical records of patients with multiple myeloma, eligible for stem cell transplantation, who received, first-line, the VTD or TD combination.

ELIGIBILITY:
Inclusion Criteria:

* clinical records of patients who were considered eligible for transplant due to their functional status and who were given some treatment strategy comprising a combination of drugs.

Exclusion Criteria:

* Incomplete clinical records
* Clinical records of patients who abandoned treatment or could not continue with the treatment due to economic or distance issues
* Clinical records of patients who presented severe sepsis before the beginning of either treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical records of patients diagnosed with multiple myeloma treated at Hospital General de México between 2020 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Favorable Response | Post-induction (6 months)
  Criteria established with the International Multiple Myeloma Working Group
Time to next treatment | Post-induction (2 years)
  Need for a secondline treatment after induction

SECONDARY OUTCOMES:
Overall survival | 3000 days
  Survivorship passing 3000 days

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo O Martinez Tovar, PhD, Study Director — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- Hospital General de Mexico Dr. Eduardo Liceaga, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
All participants and their information will be managed by intern investigators and will be kept secure for personal data protection according to Mexican laws.

REFERENCES:
- [Background] de Moraes Hungria VT, Martinez-Banos DM, Penafiel CR, Miguel CE, Vela-Ojeda J, Remaggi G, Duarte FB, Cao C, Cugliari MS, Santos T, Machnicki G, Fernandez M, Grings M, Ammann EM, Lin JH, Chen YW, Wong YN, Barreyro P. Multiple myeloma treatment patterns and clinical outcomes in the Latin America Haemato-Oncology (HOLA) Observational Study, 2008-2016. Br J Haematol. 2020 Feb;188(3):383-393. doi: 10.1111/bjh.16124. Epub 2019 Aug 7. PMID 31392724
- [Background] Mersin S, Geduk A, Mehtap O, Tarkun P, Unal S, Polat MG, Aygun K, Yenihayat EM, Albayrak H, Hacihanifioglu A. Evaluation of a Generic Bortezomib Molecule in Newly Diagnosed Multiple Myeloma Patients. Turk J Haematol. 2021 Aug 25;38(3):211-217. doi: 10.4274/tjh.galenos.2021.2020.0555. Epub 2021 May 5. PMID 33947178